CLINICAL TRIAL: NCT05011136
Title: Physician Reimbursement for Home Dialysis: Assessment of Validity of CMS Compensation for Nephrologists
Brief Title: Physician Reimbursement Home Patients
Status: Completed | Type: Observational
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: SIH 129
Record Dates: First submitted 2021-08-11; First posted 2021-08-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: ESRD
Keywords: ESRD; Home Dialysis; Compensation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. This is a qualitative study — US nephrologists who care for dialysis patients will be asked to complete an internet based survey evaluating the time and effort required for home dialysis patient care.
  Other Names: Survey

SUMMARY:
This is an observational study using an online survey to solicit information from nephrologists who care for dialysis patients about the time and effort involved in providing care to home dialysis patients.

DETAILED DESCRIPTION:
Physician reimbursement today for care of a home dialysis patient is a capitated reimbursement, defined by the age of the patient and their days on home dialysis. Due to the multiple advantages of home therapy, CMS is working on increasing home dialysis uptake; however, there is little to no data on the time and effort involved in providing care to home dialysis patients.

In this study, we will develop and distribute a survey to capture the components of home dialysis patient care and the perceived time and effort of nephrologists across the US to do so. This will provide data for CMS as they consider the adjustment of their policy values in physician reimbursement for home dialysis patient care, which is currently labeled as misvalued (Centers for Medicare and Medicaid Services, 2021).

ELIGIBILITY:
Inclusion Criteria:

* All nephrologists in the US who care for dialysis patients.

Exclusion Criteria:

* Nephrologists who have not cared for dialysis patients in the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All US nephrologists who care for dialysis patients.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To provide data to facilitate a data-driven adjustment of the capitated physician payment for caring for home dialysis patients. | Day 1
  Compilation of survey data from US nephrologists with dialysis patients.

CONTACTS AND LOCATIONS:
Overall Officials: Wael F Hussein, MBBS, Principal Investigator — Satellite Healthcare, Inc.
Locations (1):
- Satellite Health Care, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No